CLINICAL TRIAL: NCT00737724
Title: Efficacy of Simultaneous Versus Sequential Antiretroviral Therapy and Antituberculosis Treatment in Patients With AIDS and Active Tuberculosis. Open, Randomized and Controlled, Multisite Clinical Trial.
Brief Title: Simultaneous Versus Sequential Antiretroviral Therapy (ARV) Therapy and Mycobacterium Tuberculosis (MTB) Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Other published trials showed definitive expected superiority of Group 1
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Collaborators: Consorcio de Investigación sobre VIH/SIDA/TB (CISIDAT). (Other)
Responsible Party: Principal Investigator, Gustavo Reyes-Teran, Principal Investigator, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C43-06
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: HIV; AIDS; Tuberculosis
Keywords: Enzyme-Linked ImmunoSpot; Deferred treatment; Immune Recovery Inflammatory Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Antiretroviral Therapy, Highly Active; Isoniazid; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Receives both, simultaneously antiretroviral therapy and antituberculosis therapy
  Interventions: Drug: Simultaneous ARV and antiMTB
- Group 2 (Experimental): Receives only antituberculosis therapy, and 2 months afterwards antiretroviral therapy
  Interventions: Drug: Deferred RV and antiMTB treatment

INTERVENTIONS:
Drug: Simultaneous ARV and antiMTB — Receives both, simultaneously antiretroviral therapy and antituberculosis therapy
  Other Names: HAART; isoniazid; Efavirenz; Truvada
  Arms: Group 1
Drug: Deferred RV and antiMTB treatment — Receives only antituberculosis therapy and 2 months afterwards antiretroviral therapy
  Other Names: HAART; isoniazid; Efavirenz; Truvada
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate and compare the efficacy of immediate antiretroviral therapy versus 2 month deferred anti-Tb therapy upon the clinical course of tuberculosis and HIV infection in patients with AIDS and active tuberculosis.

DETAILED DESCRIPTION:
AIDS and tuberculosis are two international and national priority public health problems. The best time for starting antiretroviral therapy in patients with AIDS and active tuberculosis is not clear, despite of the guidelines regarding CD4+ count. The debate surrounding this issue is mainly due to the difficulty among adherence of anti-MTb and anti-HIV treatment, the pharmacological interaction, the adverse events related to drugs and the risk of inflammatory reconstitution syndrome, especially in patients with advanced HIV infection. Moreover, there is great debate upon the lack of knowledge of the degree of immune reconstitution throughout time against Mtb induced by the anti-HIV therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* < 200 CD4+ cells/mL
* Active pulmonary tuberculosis (with or without extrapulmonary involvement)

Exclusion Criteria:

* Meningeal tuberculosis
* Unable to attend 96 wk follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2008-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Time to remission of signs and symptoms of active tuberculosis as well as general symptoms. | 96 wk
Time to negative measurement of mycobacterial load in body fluids or affected tissues | 24 wk

SECONDARY OUTCOMES:
CD4+ cell count increase | 24 wk
Lymphoproliferative response to specific antigens against Mtb | 24 wk
Time to undetectable HIV plasma load; HIV genotype | 24 wk

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Reyes-Terán, MD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (2):
- Mexico (2):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Centro de Investigaciones en Enfermedades Infecciosas, Mexico City, Mexico City

REFERENCES:
- [Background] Raviglione MC, Narain JP, Kochi A. HIV-associated tuberculosis in developing countries: clinical features, diagnosis, and treatment. Bull World Health Organ. 1992;70(4):515-26. PMID 1394786
- [Background] De Cock KM, Soro B, Coulibaly IM, Lucas SB. Tuberculosis and HIV infection in sub-Saharan Africa. JAMA. 1992 Sep 23-30;268(12):1581-7. doi: 10.1001/jama.268.12.1581. PMID 1518113
- [Background] Whalen C, Horsburgh CR, Hom D, Lahart C, Simberkoff M, Ellner J. Accelerated course of human immunodeficiency virus infection after tuberculosis. Am J Respir Crit Care Med. 1995 Jan;151(1):129-35. doi: 10.1164/ajrccm.151.1.7812542.
- [Background] Goletti D, Weissman D, Jackson RW, Graham NM, Vlahov D, Klein RS, Munsiff SS, Ortona L, Cauda R, Fauci AS. Effect of Mycobacterium tuberculosis on HIV replication. Role of immune activation. J Immunol. 1996 Aug 1;157(3):1271-8. PMID 8757635
- [Background] Chaisson RE, Clermont HC, Holt EA, Cantave M, Johnson MP, Atkinson J, Davis H, Boulos R, Quinn TC, Halsey NA. Six-month supervised intermittent tuberculosis therapy in Haitian patients with and without HIV infection. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):1034-8. doi: 10.1164/ajrccm.154.4.8887603.
- [Background] Small PM, Schecter GF, Goodman PC, Sande MA, Chaisson RE, Hopewell PC. Treatment of tuberculosis in patients with advanced human immunodeficiency virus infection. N Engl J Med. 1991 Jan 31;324(5):289-94. doi: 10.1056/NEJM199101313240503. PMID 1898769
- [Background] Burman WJ, Jones BE. Treatment of HIV-related tuberculosis in the era of effective antiretroviral therapy. Am J Respir Crit Care Med. 2001 Jul 1;164(1):7-12. doi: 10.1164/ajrccm.164.1.2101133. No abstract available. PMID 11435232
- [Background] Dean GL, Edwards SG, Ives NJ, Matthews G, Fox EF, Navaratne L, Fisher M, Taylor GP, Miller R, Taylor CB, de Ruiter A, Pozniak AL. Treatment of tuberculosis in HIV-infected persons in the era of highly active antiretroviral therapy. AIDS. 2002 Jan 4;16(1):75-83. doi: 10.1097/00002030-200201040-00010. PMID 11741165
- [Background] Narita M, Ashkin D, Hollender ES, Pitchenik AE. Paradoxical worsening of tuberculosis following antiretroviral therapy in patients with AIDS. Am J Respir Crit Care Med. 1998 Jul;158(1):157-61. doi: 10.1164/ajrccm.158.1.9712001. PMID 9655723
- [Background] Lawn SD, Bekker LG, Wood R. How effectively does HAART restore immune responses to Mycobacterium tuberculosis? Implications for tuberculosis control. AIDS. 2005 Jul 22;19(11):1113-24. doi: 10.1097/01.aids.0000176211.08581.5a. PMID 15990564
- [Background] de Jong BC, Israelski DM, Corbett EL, Small PM. Clinical management of tuberculosis in the context of HIV infection. Annu Rev Med. 2004;55:283-301. doi: 10.1146/annurev.med.55.091902.103753. PMID 14746522
- [Background] Orlovic D, Smego RA Jr. Paradoxical tuberculous reactions in HIV-infected patients. Int J Tuberc Lung Dis. 2001 Apr;5(4):370-5. PMID 11334257
- See also: Consortium for HIV/TB Research in Mexico — http://www.cisidat.org.mx/